CLINICAL TRIAL: NCT00863980
Title: Effects of Telmisartan Compared With Candesartan on Ischemic Cardiovascular Events in High-risk Hypertensive Patients: a Multi-center, Prospective, Randomized, Open-labeled, Blinded Endpoints Trial
Brief Title: Effects of Telmisartan on Ischemic Cardiovascular Events in High-risk Hypertensive Patients
Acronym: KCPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principle investigator resigned in 2013
Sponsor: Kyoto Prefectural University of Medicine (Other)
Responsible Party: Principal Investigator, Hiroyuki Yamada, Department of Cardiovascular Medicine, Kyoto Prefectural University of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C-486; UMIN000001762
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Acute Myocardial Infarction; Angina Pectoris; Myocardial Ischemia; Acute Coronary Syndrome; Hypertension
Keywords: angiotensin; receptor; vulnerable plaque; coronary artery
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia; Acute Coronary Syndrome; Hypertension | interventions — Telmisartan; candesartan cilexetil; candesartan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telmisartan (Experimental): Treatment with Telmisartan
  Interventions: Drug: Micardis (Telmisartan)
- Candesartan (Active Comparator): Treatment with Candesartan
  Interventions: Drug: Blopress (Candesartan)

INTERVENTIONS:
Drug: Micardis (Telmisartan) — 40-80 mg/day oral administration
  Other Names: 21600AMZ00541000; Micardis Tablets 40mg
  Arms: Telmisartan
Drug: Blopress (Candesartan) — 8-12 mg/day oral administration
  Other Names: Blopless Tablets
  Arms: Candesartan

SUMMARY:
This study is aimed to investigate whether treatment with Telmisartan is more effective than Candesartan in reducing the ischemic cardiovascular events in high-risk patients with cardiovascular disease.

DETAILED DESCRIPTION:
This study is aimed to investigate whether treatment with Telmisartan is more effective than Candesartan in reducing the ischemic cardiovascular events in high-risk patients with cardiovascular disease.

Study design: PROBE(Prospective, Randomized, Open-labeled Blind Endpoints)

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are set by at least one of the three following risk factors:

1. Coronary artery disease documented by at least one of the following:

   * Myocardial infarction at least 12 months before enrollment and not planned for percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
   * Angina pectoris or asymptomatic myocardial ischemia undergoing percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) at least 12 months before enrollment and not planned for further percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
2. Peripheral arterial disease undergoing percutaneous transluminal angioplasty (PTA) or peripheral artery bypass grafting at least 6 months before enrollment
3. Symptomatic cerebral infarction or cerebral hemorrhage at least 6 months before enrollment

Exclusion Criteria:

The exclusion criteria are set as follows:

1. History of worsening of heart failure within the preceding 6 months
2. Planned elective percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within the anteceding 3 months
3. History of myocardial infarction, unstable angina pectoris, percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within the preceding 12 months
4. History of percutaneous hind limb angioplasty (PTA) or bypass grafting within the preceding 6 months
5. History of cerebral infarction, cerebral hemorrhage within the past 6 months
6. Congenital heart disease
7. Uncontrolled hypertension on treatment (eg, BP>180/110 mmHg)
8. Pregnant women or women of childbearing potential
9. Hepatic dysfunction (AST or ALT >100IU/L)
10. Renal impairment (serum creatinine level >2.0 mg per 100 ml)
11. Known hypersensitivity or intolerance to ARB

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2009-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
New or recurrent acute myocardial infarction and angina pectoris | 3 years

SECONDARY OUTCOMES:
All causes of mortality, cardiovascular death, new or recurrent stroke or peripheral artery diseases, new occurrence of diabetes mellitus | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Matsubara, MD, PhD, Study Chair — Kyoto Prefectural University of Medicine
Locations (32):
- Japan (32):
  - Shakaihoken Kobe Central Hospital, Kobe, Kobe
  - Akashi Municipal Hospital, Kobe, Kobe
  - Kouseikai Takeda Hospital, Kyoto, Kyoto
  - Aijyukai Dohjin Hospital, Kyoto, Kyoto
  - Kyoto Second Red Cross Hospital, Kyoto, Kyoto
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Social Insurance Kyoto Hospital, Kyoto, Kyoto
  - Kyoto Kojyo Hokenkai, Kyoto, Kyoto
  - Kyoto City Hospital, Kyoto, Kyoto
  - Kyoto First Red Cross Hospital, Kyoto, Kyoto
  - Aiseikai Yamashina Hospital, Kyoto, Kyoto
  - Tanabe Central Hospital, Kyoto, Kyoto
  - Rakusai Simizu Hospital, Kyoto, Kyoto
  - Uji Hospital, Kyoto, Kyoto
  - Kyoto Yawata Hospital, Kyoto, Kyoto
  - Seizinkai Simizu Hospital, Kyoto, Kyoto
  - Saiseikai Kyoto Hospital, Kyoto, Kyoto
  - Public Yamasiro Hospital, Kyoto, Kyoto
  - Gakkentoshi Hospital, Kyoto, Kyoto
  - Fukuchiyama City Hospital, Kyoto, Kyoto
  - Ayabe City Hospital, Kyoto, Kyoto
  - Maizuru Red Cross Hospital, Kyoto, Kyoto
  - National Hospital Organization Maizuru Medical Center, Kyoto, Kyoto
  - Maizuru Kyosai Hospital, Kyoto, Kyoto
  - Public Nantan Hospital, Kyoto, Kyoto
  - Kyoto Prefectural Yosanoumi Hospital, Kyoto, Kyoto
  - Kumihama Hospital, Kyoto, Kyoto
  - Sakurakai Takahashi Hospital, Kyoto, Kyoto
  - Yuuseikai Midorigaoka Hospital, Osaka, Osaka
  - Matsushita Memorial Hospital, Osaka, Osaka
  - Saiseikai Shiga Hospital, Shiga, Shiga
  - Omihachiman Community Medical Center, Shiga, Shiga